CLINICAL TRIAL: NCT01253603
Title: A Randomized, Placebo-controlled, Parallel Group Study to Assess the Efficacy, Safety, and Pharmacokinetics of QAW039 in Steroid-free Patients With Mild to Moderate Persistent Asthma
Brief Title: Efficacy, Safety, and Pharmacokinetics of QAW039
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Novartis Pharmaceuticals (Industry)
Responsible Party: Sponsor
Organization: Novartis (Industry)
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: CQAW039A2201; 2010-020177-16 (EudraCT Number)
Record Dates: First submitted 2010-12-01; First posted 2010-12-03 (Estimated); Last update posted 2020-12-19 (Actual); Status verified 2013-08

CONDITIONS: Persistent Asthma
Keywords: Asthma
MeSH Terms: conditions — Asthma | interventions — fevipiprant

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor

ARMS (3):
- 1 (Experimental): QAW039 capsules once daily for 28 days
  Interventions: Drug: QAW039 capsules once daily for 28 days
- 2 (Experimental): Placebo to QAW039 capsules once daily for 28 days
  Interventions: Drug: Placebo to QAW039 capsules once daily for 28 days
- 3 (Experimental): Fluticasone propionate inhaler twice daily for 28 days
  Interventions: Drug: Fluticasone propionate inhaler twice daily for 28 days

INTERVENTIONS:
Drug: QAW039 capsules once daily for 28 days
  Arms: 1
Drug: Placebo to QAW039 capsules once daily for 28 days
  Arms: 2
Drug: Fluticasone propionate inhaler twice daily for 28 days
  Arms: 3

SUMMARY:
This study will assess the safety, efficacy and pharmacokinetics of QAW039 in steroid-free patients with mild to moderate persistent asthma.

ELIGIBILITY:
Inclusion Criteria:

* Patients with a medical history of mild to moderate persistent allergic asthma.
* Patients must weigh at least 45 kg to participate in the study, and must have abody mass index (BMI) of >17 kg/m2.
* Female patients must be surgically sterilized, postmenopausal or using a double-barrier method of contraception

Exclusion Criteria:

* Women of child-bearing potential.
* Smokers defined as history of smoking in the previous 6 months or a smoking history of more than 10 pack years, a pack year being defined as smoking the equivalent of 20 cigarettes - a pack - every day for the period of 1 year
* Patients with severe persistent asthma

Other protocol-defined inclusion/exclusion criteria may apply.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 170 (Actual)
Dates: Start 2010-11; Primary Completion 2011-09 (Actual); Study Completion 2011-09 (Actual)

PRIMARY OUTCOMES:
Change in trough forced expiratory volume in 1 second (FEV1) compared to placebo. | 28 days

SECONDARY OUTCOMES:
To assess the safety of a 28 day administration of QAW039 compared to placebo, measured by vital signs, laboratory evaluations and electrocardiograms. | 28 days

CONTACTS AND LOCATIONS:
Overall Officials: Novartis Pharmaceuticals, Study Director — Novartis Pharmaceuticals
Locations (24):
- United States (16):
  - Novartis Investigative Site, Encinitas, California
  - Novartis Investigative Site, Huntington Beach, California
  - Novartis Investigative Site, Los Angeles, California
  - Novartis Investigative Site, Mission Viejo, California
  - Novartis Investigative Site, San Diego, California
  - Novartis Investigative Site, San Jose, California
  - Novartis Investigative Site, Stockton, California
  - Novartis Investigative Site, Stockbridge, Georgia
  - Novartis Investigative Site, North Dartmouth, Massachusetts
  - Novartis Investigative Site, Bellevue, Nebraska
  - Novartis Investigative Site, Berlin, New Jersey
  - Novartis Investigative Site, Skillman, New Jersey
  - Novartis Investigative Site, Raleigh, North Carolina
  - Novartis Investigative Site, Medford, Oregon
  - Novatis Investigative Site, Upland, Pennsylvania
  - Novartis Investigative Site, Dallas, Texas
- Novartis Investigative Site, Jambes, Belgium
- Germany (5):
  - Novartis Investigative Site, Berlin
  - Novartis Investigative Site, Cologne
  - Novartis Investigative Site, Frankfurt
  - Novartis Investigative Site, Hamburg
  - Novartis Investigative Site, Wiesbaden
- Novartis Investigative Site, Bucharest, Romania
- Novartis Investigative Site, Seoul, South Korea

REFERENCES:
- [Derived] Erpenbeck VJ, Popov TA, Miller D, Weinstein SF, Spector S, Magnusson B, Osuntokun W, Goldsmith P, Weiss M, Beier J. The oral CRTh2 antagonist QAW039 (fevipiprant): A phase II study in uncontrolled allergic asthma. Pulm Pharmacol Ther. 2016 Aug;39:54-63. doi: 10.1016/j.pupt.2016.06.005. Epub 2016 Jun 21. PMID 27354118
- See also: Results for CQAW039A2201 from the Novartis Clinical Trials website — https://www.novctrd.com/ctrdweb/trialresult/trialresults/pdf?trialResultId=10283